CLINICAL TRIAL: NCT03184051
Title: Qualification of Ultrasound Imaging Technique in the Quantitative Evaluation of Cartilaginous Tissue of Femoral Condyle Articulation and Osteoarthritis
Brief Title: Diagnostic Performance of Ultrasound Imaging Technique for Femoral Condyle Cartilage Evaluation and Osteoarthritis
Acronym: CARTILAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: 38RC17.074
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Ultrasonography evaluation/ultrasound; Articular cartilage; UltraSound Speed Of Sound (US-SOS); UltraSound Time of Flight (US-TOF)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound assessment: All subject of the study have a knee osteoarthritis (OA) and are going to have a total arthroplasty. Diagnostic performance of ultrasonography is evaluated on ex vivo cartilage samples (2 samples per patient are selected with different stage of OA : 1 with early stage and 1 with advanced stage).

SUMMARY:
This study investigates the potential of the ultrasound imaging technique to diagnose the severity of knee osteoarthritis (OA). In parallel, measurements will also be conducted using Magnetic Resonance Imaging (MRI) and histology analysis as reference tools.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a common degenerative disease of synovial joint becoming more frequent with age. Among techniques have been used to diagnose and classify the severity of knee OA, the imaging techniques, such as ultrasonography (US), provide physical quantitative informations for better understanding and assessing of the pathology of the knee joint.

The present study aim to investigate the diagnostic performance of ultrasonography for femoral condyle cartilage evaluation using MRI and histology analysis as reference tools. To validate this approach, evaluations are conducted to determine, whether the UltraSound Speed Of Sound (US-SOS) propagation is associated with the variation of the arthrosis stage, in order to improve the diagnosis of the surgeon. For this purpose, measurements are conducted using selected human cartilage samples with different stage of OA (early stage and advanced stage).

This research is the first "preclinical" study of a new unlabelled medical device developed by Cartimage Medical SAS. Cartilage is a prospective, monocentric, unrandomized and uncontrolled study. This study doesn't modify the medical care of the patient.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 year old
* knee osteoarthritis which total knee arthroplasty indication
* who have signed a non-objection form.

Exclusion Criteria:

* person who refuse to sign a non-objection form
* person deprived of liberty by judicial or administrative decision
* person under legal protection or unable to express their consent
* person hospitalized for psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis with an indication of total arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the correlation between the Time of Flight (TOF) of ultrasounds between the two interfaces (bone / cartilage and cartilage / water) and the real thickness of the cartilage measured by Magnetic Resonance Imaging (MRI). | 5 months
  Correlation coefficients between US-TOF measurements and cartilage thickness measurements corresponding to MRI.

SECONDARY OUTCOMES:
Evaluation of the relationship between the propagation velocity of the ultrasound wave in cartilage tissue and the osteoarthritis degree defined by OARSI scale. | 5 months
  Correlation coefficients between the US propagation velocity measurements and OA progression according to the seven groups of the OARSI scale.
  Position indicators of US propagation velocity measurements of the 2 groups "early stage" (0 <= OARSI <= 2) and "advanced stage" (3 <= OARSI <= 6).
Evaluation of the relationship between 3D surface reconstruction and defects of cartilage samples from localized ultrasound data and those derived from MRI data | 5 months
  Correlation coefficient between surface area of samples and defects estimated from ultrasound data and those derived from MRI data.
  Correlation coefficients between surface volumes of samples and defects estimated from ultrasound data and those derived from MRI data.
Evaluation of correlation between thickness measured by MRI and this measured by histological analysis. | 5 months
  Correlation coefficients between thickness measurements estimated from MRI data and those estimated from histological data.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau -Gaudry, MD, PhD, Principal Investigator — Clinical Investigation Centre for Innovative Technology Network - University Hospital Grenoble
Locations (1):
- Orthopedic Surgery Department, University Hospital, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description: Clinical Investigation Centre for Innovative Technology Network website — http://www.cic-it.fr/cic-it-grenoble.php